CLINICAL TRIAL: NCT04689126
Title: Effect of Cone Beam Computed Tomography on Diagnostic and Therapeutic Decision Making in Endodontics
Brief Title: Effect of Cone Beam Computed Tomography on Diagnostic and Therapeutic Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: natwar singh
Record Dates: First submitted 2020-12-11; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Diagnoses Disease
Keywords: resorption; fracture; pulp necrosis; nonendodontic diagnosis
MeSH Terms: conditions — Fractures, Bone; Dental Pulp Necrosis | interventions — Surgical Procedures, Operative; Apicoectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention (Experimental): diagnosis and treatment plan before and after cone beam computed tomography scan
  Interventions: Procedure: surgical or nonsurgical endodontic treatment

INTERVENTIONS:
Procedure: surgical or nonsurgical endodontic treatment — Change in diagnosis and treatment plans between the two imaging - periapical radiography and cone beam computed tomography
  Other Names: extraction; root amputation

SUMMARY:
this study will determine the effect of CBCT examinations on diagnostic and therapeutic decision making in endodontics.

DETAILED DESCRIPTION:
Patients selected for Cone beam computed tomography (CBCT) examinations in accordance with European Commission guidelines ( patients with symptomatic vital teeth or with symptomatic root filled teeth; patients with suspected dental fracture; patients with suspected external or internal resorption and for aid in performing any therapeutic intervention ) will be included in the study. Only patients aged above 18 years will be included in the study.

Patients referred to the department of endodontics at Post Graduate Institute of Dental Sciences (PGIDS) Rohtak or any patient from routine opd requiring specialist endodontic consultation will be thoroughly examined .The examination will consist of a proper medical history and clinical examination, such as inspection, palpation, probing and percussion of the area of interest. When appropriate, additional tests such as sensitivity tests (cold and electric pulp tests) and conventional radiography will be performed. After the initial examination, patients judged to be in need of CBCT examination will be referred to the radiology department.

Stages of evaluation

Stage 1(before CBCT examination) Before referral, the examiner will write down the best available diagnosis and therapeutic plan using clinical examination and conventional radiography. The radiographs will be carefully viewed for periapical changes, vertical root fractures, internal or external resorption, perforation or any other radiographic finding.

Stage 2(after CBCT examination)

After the CBCT examination, the previous diagnosis and treatment plan will be considered and, if needed, a new diagnosis and treatment plan will be made by the same examiner, taking into consideration all of the data. The examiners will have access to all image reconstructions performed by the radiologist. These reconstructions will include images in the axial, coronal and sagittal planes throughout the entire volume.

Stage 3(patient dismissal) As per requirement therapy will be performed on the patients. The findings of orthograde treatment, explorative surgery, endodontic microsurgery, or extraction will serve as a gold standard for definitive clinical diagnosis.

Radiological investigation All intraoral periapical radiographs will be done with at least two angled (mesial and distal) views.

CBCT examination (Kodak CS 9300 Care Stream) done with exposure parameters 85 kilovolt and 5ma isotropic voxels with a size of 90*90*90 microns 5 *5 cm volume FOV Slice thickness will vary from .9 to 1.3 mm.

The images will be viewed on a screen with a resolution of 1280*1024pixels (Dell E19135).

Diagnostic decision making The diagnosis with periapical radiograph and CBCT will be made as per following choices

1. Healthy
2. Pulp necrosis
3. Apical periodontitis
4. External resorption
5. Root fracture
6. Non-endodontic diagnosis
7. Others

Therapeutic decision making

Treatment plans decided by radiographs and CBCT will be divided into following choices

1. No treatment
2. Wait and watch
3. Orthograde endodontics
4. Retrograde endodontics
5. Explorative surgery
6. Extraction
7. Referral to other specialist
8. Others

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for referring patients to CBCT examination will be in accordance with current European guidelines and can be grouped as follows:

  1. Patients in which disease had to be ruled out:

     1. patients with symptomatic vital teeth otherwise judged healthy (no exposed dentin; normal sensitivity pulp tests; no tenderness to palpation or percussion; with radiographic apical/marginal periodontal normalcy; and no cracks/fractures)
     2. patients with symptomatic root-filled teeth otherwise judged healthy (good quality of root filling that did not need to be revised or completed; no tenderness to palpation or percussion; with radiographic apical/marginal periodontal normalcy; and no cracks/fractures)
     3. when conventional radiology failed to demonstrate if a finding was a pathological process or a normal anatomical structure.
  2. Patients in which suspected disease had to be confirmed:

     1. suspected dental fractures that could not be demonstrated
     2. suspected external or internal resorptions.
  3. As an aid in performing the therapeutic intervention:

     1. in established external or internal resorptions to assist in the approach of complex cases
     2. before apical surgery when important anatomical structures interfered with the surgical approach
     3. in diagnosing foreign body structures, their location and, when needed, as a guide in the surgical removal
     4. in understanding tooth anatomy of abnormal teeth in need of endodontic treatment
     5. in assessing the number and location of root canals after at least one unsuccessful attempt to find them under oral microscope.

Exclusion Criteria:

* Patients will not be referred for CBCT examination if they:

  1. presented themselves with an accessible previous volume tomography in the region of interest. This was, however, not a strict restriction if the examiner judged that new and relevant information could be obtained by a new CBCT examination
  2. had a definite diagnosis and treatment plan after a complete clinical and conventional radiographic examination and therefore did not need a CBCT examination. This group represented the vast majority of all patients
  3. needed any other special imaging technique for soft tissue assessment such as CT or magnetic resonanace imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in diagnosis and treatment planning | 1 year
  Comparison of diagnostic and therapeutic decision making between gold standard and radiographic findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Science, Rohtak, Haryana, India